CLINICAL TRIAL: NCT04001361
Title: Combined Effect of IPG Medical Charlie Laser and Bone Marrow Grafting on Cartilage Defects of the Knee
Brief Title: Laser Cell Therapy for Knee Cartilage Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Endocellutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LRK1
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Blinded trial. Three groups. Sham, laser only, laser plus marrow. Stage 2 and 3 OA of one or both knees
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sham laser means laser not turned on. Sham marrow means incision in skin made but no marrow drawn. Patient under conscience sedation. MRI and outcomes measures independently measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham (Sham Comparator): Under conscience sedation, a nick in the skin is made to mimic marrow aspiration. Laser inserted into knee joint but not turned on.
  Interventions: Procedure: Laser Cell Therapy
- Laser Only (Experimental): Under conscience sedation, a nick in the skin is made to mimic marrow aspiration. Laser fiber is inserted into knee over an 18 gauge needle and micro-channels are made into the damaged cartilage.
  Interventions: Procedure: Laser Cell Therapy
- Laser plus Marrow (Experimental): Under conscience sedation, a 10mL marrow aspiration is performed. Laser fiber is inserted into the knee over an 18 gauge needle and micro-channels are made into the damaged cartilage. After the channels are made, marrow aspirate is injected over the same 18 gauge needle.
  Interventions: Procedure: Laser Cell Therapy

INTERVENTIONS:
Procedure: Laser Cell Therapy — Bone marrow aspirate combined with laser to alter the cartilage matrix to facilitate repair

SUMMARY:
Laser pulsed energy will be delivered over an optical fiber to create channels into damaged cartilage of the knee or knees. The channels have a diameter of approximately 100 microns or less and an approximate depth of 1 millimeter or less. Bone marrow aspirate will then be delivered into the damaged joint.

DETAILED DESCRIPTION:
The creation of micro-channels into damaged knee cartilage will facilitate the movement of fluid into and out of the tissue to allow for more efficient nutrient diffusion. The addition of bone marrow aspirate will provide additional growth factor enriched nutrition to the tissue. The goal of this combination therapy is to facilitates the body's own reparative processes leading to improved patient well being.

ELIGIBILITY:
Inclusion Criteria:

Kellergren grading scale of 2 or 3 in at least one compartment of either or both knees with no compartment representing a stage 4 in either knee.

No significant MCL or LCL tear or laxity

No significant meniscal tear. ( i.e. bucket handle)

Exclusion Criteria:

* Injection with the past 6 weeks
* Stage 4 osteoarthritis in either knee
* Uncontrolled Diabetes or any other metabolic syndrome
* BMI greater than 28
* Significant lower extremity deformity
* Bilateral or tri compartmental Knee OA
* Adults unable to consent
* Individuals who are not yet adults (infants, children, and teenagers, age < 18)
* pregnant women
* Prisoners
* Stage 4 osteoarthritis in either knee
* Subjects, who, in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI | one year
  Pre procedure MRI and post MRI is taken to measure disease modification
VAS Score | one year
  Pre procedure and post procedure Pain score
KOOS score | one year
  Pre procedure and post procedure Improvement in daily living and pain
Treadmill Test | one year
  Pre procedure and post procedure, the patient will walk for 12 minutes with a gradual increase and a change in pain will be evaluated
Swiss Ball wall squat test | one year
  Swiss Ball wall squat test to asses functional recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scarpone, Principal Investigator — Trinity Sports Medicine
Locations (1):
- Trinity Sports Medicine, Steubenville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared unless the principal investigator decides to make public either through podium presentations or written publication.